CLINICAL TRIAL: NCT07025577
Title: A Phase 1, Open-Label, Fixed-Sequence, Randomized Study to Assess the Tolerability and Safety of Subcutaneously Administered Immunoglobulin G With Varying Injection Conditions
Brief Title: A Study to Assess the Tolerability and Safety of Subcutaneously (SC) Administered Immunoglobulin G (IgG) With Varying Injection Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP45580
Record Dates: First submitted 2025-05-30; First posted 2025-06-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Participants will receive SC administrations of IgG into the abdominal region starting with Treatment B, followed by Treatment A.
  Interventions: Drug: Immunoglobulin G
- Sequence 2 (Experimental): Participants will receive SC administrations of IgG into the abdominal region starting with Treatment A, followed by Treatment C.
  Interventions: Drug: Immunoglobulin G
- Sequence 3 (Experimental): Participants will receive SC administrations of IgG into the abdominal region starting with Treatment D, followed by Treatment C.
  Interventions: Drug: Immunoglobulin G
- Sequence 4 (Experimental): Participants will receive SC administrations of IgG into the abdominal region starting with Treatment B, followed by Treatment D.
  Interventions: Drug: Immunoglobulin G

INTERVENTIONS:
Drug: Immunoglobulin G — Participants will receive SC administrations of IgG

SUMMARY:
This study will evaluate the safety and tolerability of SC administration of IgG in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 36 kilograms per meter square (kg/m^2), inclusive
* For females of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during IgG administration and for 28 days after completion of IgG administration
* For males: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 28 days after the last study drug administration
* Positive human immunodeficiency virus (HIV) test
* Positive hepatitis B surface antigen or hepatitis B core antibody test
* Positive hepatitis C virus antibody test
* Regular alcohol consumption of >8 drinks/week for females or >12 drinks/week for males
* Poor peripheral venous access
* Major surgical procedure within 28 days prior to initiation of study treatment or anticipation of need for a major surgical procedure during the study
* Known hypersensitivity to IgG or any of its components or to products made with IgG
* History or presence of skin rash or other skin disorders
* Inability to sense pain (e.g., peripheral neuropathy) or have a history of or have been diagnosed with a chronic pain syndrome
* Infection or inflammation of the designated injection site (abdomen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Mean Injection Site Tolerability Score on a Visual Analogue Scale (VAS) | Up to Day 4
Mean Change From Baseline in Injection Site Tolerability Score on VAS | Baseline, Up to Day 4
Percentage of Participants Experiencing Greater Than Mild Pain | Up to Day 4
Percentage of Participants in Each VDS Category on the VDS Scale | Up to Day 4
Percentage of Participants with Local Injection Site Reaction Using Local Injection-site Symptom Assessment (LISSA) | Up to Day 7
Participant's Tolerability to Injection as Assessed by Tolerability Questionnaire | Up to Day 4
Number of Participants with Visual Injection Site Tolerability as assessed using LISSA | Up to Day 4
Number of Participants with Fluid Leakage | Up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Daytona Beach Clinical Rsch Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas
  - Fortrea Clinical Research Unit Inc. - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No